CLINICAL TRIAL: NCT02161939
Title: A Multicenter Treatment Protocol of Daclatasvir (BMS-790052) in Combination With Sofosbuvir for the Treatment of Subjects With Chronic Hepatitis C and Decompensated Cirrhosis or Post-Liver Transplant Subjects With Chronic Hepatitis C Recurrence
Brief Title: A Multicenter Treatment Protocol of Daclatasvir (BMS-790052) in Combination With Sofosbuvir for the Treatment of Post-Liver Transplant Subjects With Chronic Hepatitis C
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-257
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; Sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir (BMS-790052)
Drug: Sofosbuvir

SUMMARY:
The primary objective of this program is to provide DCV for 24 weeks to be given in combination with SOF to subjects with chronic hepatitis C with decompensated cirrhosis or post-liver transplant subjects with chronic hepatitis C recurrence with either advanced fibrosis or fibrosing cholestatic hepatitis and who have a serious or immediately life-threatening condition or experienced an event that has decreased their life expectancy to <12 months, therefore, no research hypothesis will be tested and no specific endpoints are defined. However, safety data will be collected throughout the study as well as efficacy data

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients chronically infected with Hepatitis C
* Subjects who received a liver transplant, have chronic hepatitis C virus (HCV) recurrence and advanced fibrosis (Metavir F3-F4) or fibrosing cholestatic hepatitis
* Subjects with decompensated cirrhosis defined by Child-Pugh Class C

Exclusion Criteria:

* Patients who are <18 years old
* Clinical or pathologic evidence of acute ongoing liver graft rejection
* Creatinine clearance (CrCl) ≤30 mL/min (as estimated by Cockcroft and Gault formula)
* Patients who have contraindications to either Daclatasvir (DCV) or Sofosbuvir (SOF)
* Patients who are pregnant or Women of Child Bearing Potential who are not using required contraception

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (20):
  - Mayo Clinic, Phoenix, Arizona
  - USC - Keck Medical Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Piedmont Transplant, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - Mass General, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, University Campus, Worchester, Massachusetts
  - Henry Ford, Detroit, Michigan
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC, Chapel Hill, North Carolina
  - Carolinas Healthcare Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadephia, Pennsylvania
  - Research Specialist of Texas, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Hospital, Seattle, Washington

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx